CLINICAL TRIAL: NCT00212004
Title: The Japan Working Group for the Assessment That the Pioglitazone Protects DM Patients Against Re-Infarction
Brief Title: Pioglitazone Protects Diabetes Mellitus (DM) Patients Against Re-Infarction (PPAR Study)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Limited budget to continue this study
Sponsor: National Cerebral and Cardiovascular Center, Japan (Other)
Collaborators: Japan Heart Foundation (Other)
Responsible Party: Principal Investigator, Masafumi Kitakaze, Department of Clinical Medicine and Development, National Cerebral and Cardiovascular Center, Japan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CSSCJ-4; UMIN_ID:C000000091; Umin Center (Other: Japanese government)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Diabetes Mellitus; Myocardial Infarction
Keywords: diabetes mellitus; myocardial infarction; pioglitazone
MeSH Terms: conditions — Diabetes Mellitus; Myocardial Infarction | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pioglitazone (Active Comparator): Participants in the pioglitazone group were administered a pioglitazone tablet (15 mg) once a day. In the event of the side effects such as oedema, the dosage of pioglitazone was reduced to half or a quarter of the original dosage. Otherwise, we tried to increase the dose of pioglitazone to 30mg/day.
  Interventions: Drug: pioglitazone
- Control (Active Comparator): Participants assigned to Control group were treated with diet and exercise therapy or sulfonylurea (SU) or other additional drugs than pioglitazone.
  Interventions: Other: control

INTERVENTIONS:
Drug: pioglitazone
  Arms: Pioglitazone
Other: control
  Arms: Control

SUMMARY:
To evaluate whether the pioglitazone could reduce the recurrence of myocardial infarction (MI) in patients with DM and old myocardial infarction

DETAILED DESCRIPTION:
Type 2 diabetes mellitus is a well-established risk factor for coronary heart disease and atherosclerotic change in coronary artery. So we designed a prospective randomized multi-center trial named the pioglitazone could reduce the recurrence of myocardial infarction in patients with DM and myocardial infarction(PPAR study) to evaluate whether pioglitazone could reduce the recurrence of myocardial infarction in patients with DM(HbA1c<6.5%) and myocardial infarction.

More than 100 hospitals will participate in the PPAR study. Patients with DM who have history of prior myocardial infarction are randomly allocated to receive pioglitazone or (1)instructs weight reduction, appropriate diet, regular exercise and/or (2)prescribes sulfonylurea agents. The number of patients to be recruited is 720 and this study will continue at least 2 years until 7 year or the end of the study. The primary end-points are (1) cardiovascular mortality and (2) hospitalization for cardiovascular events. Effects in suppression of new diabetes development also will be evaluated.

We should recognize DM as important therapeutic target to decrease recurrence of cardiovascular events. PPAR study, a large scale multi-center trial in Japan, will provide us new evidence how to treat DM patients with prior myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

1. diabetes mellitus (fasting plasma glucose levels of>126 mg/dL, or 2-hour 75g oral glucose tolerance test (OGTT) value of >200 mg/dL, and HbA1c levels of<6.5% (47.5 IFCC))
2. History of myocardial infarction
3. Age between 20-79 years old

Exclusion Criteria:

1. acute MI occurring within the last 7 days
2. New York Heart Association (NYHA) symptoms of no fewer II or with left ventricular ejection fraction of not more than 40%
3. suspected type I DM
4. scheduled coronary angioplasty or history of coronary artery bypass graft surgery
5. serious liver or kidney damage
6. history of allergy or drug hypersensitivity
7. arteriosclerosis obliterans with Fontaine stage III or worse
8. inability to understand and/or comply with study medications, procedures and/or follow-up or any conditions that may render the patient unable to complete the study in the opinion of the investigator.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Actual)
Dates: Start 2005-04 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
The time till the first cardiovascular composite endpoint | 2 years
  death from cardiovascular death, and the hospitalization due to nonfatal myocardial infarction, nonfatal unstable angina25, treatment with coronary revascularisation (percutaneous coronary intervention or coronary artery bypass graft) and cerebral infarction.

SECONDARY OUTCOMES:
All cause mortality | 2 years
  death of any cause
Hospitalization due to nonfatal myocardial infarction | 2 years
  nonfatal myocardial infarction
Hospitalization due to nonfatal unstable angina | 2 years
  nonfatal unstable angina
Hospitalization due to treatment with coronary revascularisation (percutaneous coronary intervention or coronary artery bypass graft) | 2 years
  coronary revascularisation
Hospitalization due to cerebral infarction | 2 years
  cerebral infarction
The progression of DM | 2 years
  HbA1C levels>7.0%
worsening of renal function | 2 years
  serum creatine levels>2.5mg/dL or the increases of serum creatine levels by >2mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Masafumi Kitakaze, MD, PhD, Study Chair — National Cerebral and Cardiovascular Center, Japan
Locations (1):
- National Cardiovascular Center, Suita, Osaka, Japan